CLINICAL TRIAL: NCT01400854
Title: ERKENTNIS: Effentora® in Clinical Practice - a Non-interventional Study to Evaluate Satisfaction and Tolerability
Brief Title: Effentora® in Clinical Practice - a Non-interventional Study to Evaluate Satisfaction and Tolerability
Acronym: ERKENTNIS
Status: Completed | Type: Observational
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: C25608/5008
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Cancer; Pain
Keywords: breakthrough cancer pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Effentora®: Single group prospective treatment cohort
  Interventions: Drug: Effentora®

INTERVENTIONS:
Drug: Effentora® — prescribed as per local Summary of Product Characteristics (SmPC) for 4 weeks duration

SUMMARY:
Aim of this non-interventional study is to investigate the tolerability of Effentora® in cancer pain patients with breakthrough pain under real-life conditions in clinical practice.

DETAILED DESCRIPTION:
In addition to the effectiveness of Effentora® therapy, safety, general feasibility and the impact of therapy on the patients' quality of life are of interest.

ELIGIBILITY:
Inclusion Criteria:

* decision to start treatment with Effentora
* prescription in accordance with Summary of Product Characteristics (SmPC)
* personally signed and dated Informed Consent document

Exclusion Criteria:

* any subject considered unsuitable according to SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients (in- or out-patients) that are suffering from breakthrough pain
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
pain relief | 4 weeks
  to show adequate pain relief within 10 minutes

SECONDARY OUTCOMES:
occurrence of adverse events | 4 weeks
  document the tolerability of Effentora®
Change in level of breakthrough pain | 4 weeks
  pursue the possible changes in the history of breakthrough pain during treatment with Effentora
presence of specific triggers for breakthrough pain | 4 weeks
  to investigate the presence of specific triggers (directly or indirectly) with breakthrough pain
quality of life | 4 weeks
  to document the impact of breakthrough pain in different areas of patients' lives and their changes during treatment with Effentora®

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Cephalon
Locations (1):
- Cephalon GmbH, Munich, Bavaria, Germany